CLINICAL TRIAL: NCT01698086
Title: Vestibular Rehabilitation for Persons With Multiple Sclerosis: Who Benefits the Most?
Brief Title: Vestibular Rehabilitation for Persons With Multiple Sclerosis: Who Benefits the Most? (MSVR3trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-1114; RG 4710A1/1 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis; Balance; Fatigue; Eye Movement
Keywords: Multiple Sclerosis; Balance; Fatigue; Eye movement
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Participants who are randomized to the Experimental group will perform 1-hour supervised intervention sessions 2x/wk for 6-wks, then 1x/wk for 8-weeks, for a total of 20 supervised sessions (Figure 1). The intervention is a progressive vestibular rehabilitation program comprised of balance and eye movement exercises as detailed in our preliminary study report.
  Interventions: Other: Vestibular rehabilitation: balance and eye movement exercises
- Wait-listed Control group (No Intervention): The Wait-listed Control group will not receive treatment; however, participants in the Wait-listed Control group will undergo the same outcome measurement plan as the Experimental group. If interested, participants from this group will be placed on a wait-list and will have the opportunity to receive instructions in how to perform the vestibular rehabilitation program following their completion of the study.

INTERVENTIONS:
Other: Vestibular rehabilitation: balance and eye movement exercises — The Experimental group will perform 1-hour supervised intervention sessions 2x/wk for 6-wks, then 1x/wk for 8-weeks, for a total of 20 supervised sessions. The intervention is a progressive vestibular rehabilitation program comprised of balance and eye movement exercises as detailed in our preliminary study report. The balance training includes standing and walking tasks on varied types of compliant surfaces, base of support, head movements, visual input and eye-hand tasks. The tasks will progress from simple to more complex. Eye movement exercises will include voluntary saccadic eye movements and smooth pursuit movements. Vestibulo-ocular eye training will be performed while visually fixating on a stationary object, while moving the head up and down and side to side at various speeds, progressing from sitting to standing on firm and compliant surface. Participants in the Experimental group will be given items of the exercise program to perform as a home exercise program.
  Arms: Experimental group

SUMMARY:
Impaired standing balance, fatigue and abnormal eye movements are common problems in persons with MS. These complaints are related to advanced disability and decreased quality of life for persons with MS. Researchers from the University of Colorado and the Rocky Mountain Multiple Sclerosis Center (RMMSC) at the Anschutz Medical Campus have recently completed and published a research study that showed an exercise program consisting of balance and eye movement training, referred to as a vestibular rehabilitation program, was very effective in improving self-reported fatigue and standing balance in persons with MS. This initial study was the first to have proven that this type of exercise program is able to improve both of these potentially devastating complaints.

The investigators from this initial study have partnered with other well-established researchers from the University of Colorado Anschutz Medical Campus and the Rocky Mountain Multiple Sclerosis Center (RMMSC) at the Anschutz Medical Campus to advance our knowledge of the effect of vestibular rehabilitation for persons with MS. Using the findings from the initial study, the investigators propose to conduct a larger study specifically identifying persons with MS who have brain lesion involvement in areas that control balance and eye movements. Primarily, the current study will determine if those individuals who have involvement in these areas of the brain improve more in balance and fatigue compared to those who do not following participation in a vestibular rehabilitation program. Additionally, the investigators will test if study participants who have abnormal eye movement control, will improve their eye movement control following the training program. For persons with MS, impaired eye movements can lead to a considerable decline in health status, further illustrating the importance of the research plan to study this important factor.

The investigators believe that greater improvements in balance and fatigue are possible from a longer treatment, and that participants who have brain lesion involvement in areas that help control balance and eye movements will benefit greater than those who do not. This information is important to determine who is more likely to benefit from a vestibular rehabilitation program. Additionally, the researchers will be able to measure changes in eye movement control, providing valuable insight into the reasons for the program's effectiveness.

DETAILED DESCRIPTION:
Hypotheses and Specific Aims

Specific Aims Impaired balance (upright postural control), visual instability and fatigue are common complaints in persons with multiple sclerosis (MS), often leading to advanced disability and lower quality of life. MS affects structures throughout the central nervous system (CNS), with frequent involvement of infratentorial structures including the brainstem and cerebellum.1-4 These structures play integral roles in the process of maintaining balance.5-8 Indeed, for the person with MS, involvement of these structures is strongly linked to impaired balance, often leading to falls.9,10 To our knowledge, no studies have established effective treatment to improve balance specifically for persons with MS who have involvement of brainstem/cerebellar structures.

Our previous study11 provides evidence that vestibular rehabilitation, an exercise program involving balance and eye movement training, greatly improves balance and fatigue in patients with MS who have primary complaints in these areas. Brainstem and cerebellar dysfunctions are strongly associated with impaired balance.9,10 Analysis from our previous study indicates that greater improvements in balance from vestibular rehabilitation are likely for persons with MS who have brainstem and/or cerebellar involvement. Neural plasticity has been reported in persons with MS following task-specific training.12-15 We conceptualize that vestibular rehabilitation targets the CNS, specifically the brainstem and cerebellum, by providing the necessary task-specific stimuli for effective neural reorganization, improving central sensory integration resulting in improved balance and visual stability. Functioning with impaired balance and visual stability can be highly fatiguing. As such, we anticipate that this intervention approach also improves fatigue.

We propose a 16-wk, two-group, stratified-blocked randomized controlled trial. Our primary aim is to determine if vestibular rehabilitation for persons with MS is more effective in improving balance for those who have brainstem and/or cerebellar involvement compared to persons with MS who do not. In addition, because eye movement exercises are an important part of the proposed vestibular rehabilitation program, we will determine if significant changes in visual stability for persons with MS who present with abnormal eye movements are possible following participation in this program. Lastly, we will expand our knowledge of the benefits of vestibular rehabilitation on fatigue

Primary Aim: To compare changes in balance based on two strata: participants with brainstem and/or cerebellar involvement and those without, and to compare changes between the two study groups: Experimental group (vestibular rehabilitation program) and Wait-listed Control group (wait-listed for vestibular rehabilitation instruction).

Hypothesis (H1): 1) Participants in the Experimental group having brainstem and/or cerebellar involvement will have greater improvements in balance compared to those without brainstem and/or cerebellar involvement; 2) The Experimental group will have greater improvements in balance compared to the Wait-listed Control group.

Secondary Aim 1: To identify changes in eye movement dysfunction for participants in the Experimental group having eye movement dysfunction at baseline, and to compare changes between the two study groups.

Hypothesis (H2): 1) Participants in the Experimental group who present with impaired eye movements at baseline will improve significantly in visual stability following performance in the vestibular rehabilitation program compared to baseline values; 2) Participants in the Experimental group who present with impaired eye movements will improve significantly in visual stability compared to participants in the Wait-listed Control group who also present with impaired eye movements.

Secondary Aim 2: To compare changes in self-reported fatigue based on brainstem and/or cerebellar involvement stratum and between the two study groups.

Hypothesis (H3): 1) Participants in the Experimental group having brainstem and/or cerebellar involvement will have greater improvements in fatigue compared to those without brainstem and/or cerebellar involvement; 2) The Experimental group will have greater improvements in fatigue compared to the Wait-listed Control group.

An overarching objective of our research is to set the stage for future investigations of the underlying mechanisms responsible for the benefits found from vestibular rehabilitation. CNS involvement and neural plasticity will serve as primary targets of future investigations.

ELIGIBILITY:
Inclusion Criteria:

* clinically definite MS confirmed by a neurologist
* walk 100 meters with no greater than intermittent or unilateral constant assistive device support (coinciding with a Kurtzke Expanded Disability Status Scale (EDSS) range of 1.0 to 6.0: 1.0 to 4.5 fully ambulatory without assistive device; 5.0 to 5.5 impaired ambulatory status without assistive device; 6.0 impaired ambulatory status with intermittent or unilateral constant assistive)
* 18 to 60 years of age
* able to speak, read and understand English
* provide informed consent
* report at least a moderate level of fatigue (MFIS total score > 22)
* at least moderate level of impaired balance (SOT composite score < 82)
* minimal leg spasticity: score of <1 for the legs on the Modified Ashworth spasticity scale (score range: 0 - 4; 0 indicates no spasticity present, 4 is legs are rigid in all directions; 1 = indicates slight increased muscle tone)

Exclusion Criteria:

* non-ambulatory
* use of unilateral or bilateral foot, ankle and/or knee orthoses.
* medical history of other possible causes of fatigue (e.g. major sleep disorder, clinically diagnosed major depressive disorder, anemia, hypothyroidism, B12 deficiency, cancer)
* complete or legal blindness in one or both eyes.
* neurological disorder which might contribute to significant balance problems, such as cerebral vascular accident, peripheral neuropathy (including diabetes mellitus), peripheral vestibular disorders (unilateral/bilateral vestibular hypofunction: benign positional paroxysmal vertigo, Meniere's disease, acoustic neuroma)
* documented MS-related exacerbation in the last three months.
* medical diagnosis or condition (e.g. cardiac, pulmonary, hepatic) that is considered to be an absolute or relative contraindication to participating in exercise
* participation in an exercise routine specifically designed to improve balance, fatigue and/or visual stability within 12 weeks prior to study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Balance (Dynamic Posturography/Computerized Sensory Organization Test) | 6 weeks and 14 weeks
  Change in balance from Baseline to 6 weeks and 14 weeks

SECONDARY OUTCOMES:
Visual Stability (Dynamic Visual Acuity and Gaze Stabilization Test) | 6 weeks and 14 weeks
  Change from Baseline in Visual Stability at 6 weeks 14 weeks
Perceived fatigue (Modified Fatigue Impact Scale) | 6 weeks and 14 weeks
  Change from Baseline in Perceived fatigue at 6 weeks 14 weeks.

OTHER OUTCOMES:
Disability due to dizziness or disequilibrium (Dizziness Handicap Inventory) | 6 weeks and 14 weeks
  Change from Baseline in Disability due to dizziness or disequilibrium at 6 weeks 14 weeks.
Change in Walk Speed (Timed 25 Foot Walk Test) | 6 weeks and 14 weeks
  Change from Baseline in Walk Speed at 6 weeks and at 14 weeks.
Change in Health Status (SF-36) | 6 weeks and 14 weeks
  Change from Baseline in Health Status at 6 weeks and at 14 weeks.
Cognition (Perceived Deficits Questionnaire) | 6 weeks and 14 weeks
  Change from Baseline in Cognition at 6 weeks and 14 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Hebert, PhD, PT, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus/University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Hebert JR, Corboy JR, Vollmer T, Forster JE, Schenkman M. Efficacy of Balance and Eye-Movement Exercises for Persons With Multiple Sclerosis (BEEMS). Neurology. 2018 Feb 27;90(9):e797-e807. doi: 10.1212/WNL.0000000000005013. Epub 2018 Jan 31. PMID 29386274